CLINICAL TRIAL: NCT01845220
Title: Prevention of Alcohol Intolerance
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00081276
Record Dates: First submitted 2013-04-23; First posted 2013-05-03 (Estimated); Results first posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-08

CONDITIONS: Alcohol Sensitivity
Keywords: Broccoli sprouts; alcohol sensitivity; sulforaphane; alcohol metabolism; in the Asian Community

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Broccoli Sprout Extract (Active Comparator): Each subject will act as his/her own control and receive both treatment and placebo on adjacent skin regions.
  Interventions: Drug: Broccoli Sprout Extract
- Placebo (Placebo Comparator): Each subject will act as his/her own control and receive both treatment and placebo on adjacent skin regions.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Broccoli Sprout Extract — 150 nanomol of sulforaphane/cm2 of skin in 80% acetone for 3 applications on 3 successive days prior to alcohol challenge
  Arms: Broccoli Sprout Extract
Drug: Placebo — 80% acetone
  Arms: Placebo

SUMMARY:
This study is designed to determine whether Asians who are especially sensitive to alcohol exposure can be protected by boosting their activities of an alcohol disposing enzyme. This will be accomplished by administering broccoli sprouts that are rich in an agent that increases protective enzyme activity. The test system involves applying alcohol patches to the skin and measuring skin redness.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years old,
* sensitive to alcohol on the skin, Japanese

Exclusion Criteria:

* recent skin abnormalities /tanning

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07-01 (Actual); Study Completion 2015-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: skin area
Period: Overall Study
Arm/Group | Broccoli Sprout Extract | Placebo
Started | 30; 30 skin area | 30; 30 skin area
Completed | 30; 30 skin area | 30; 30 skin area
Not Completed | 0; 0 skin area | 0; 0 skin area

BASELINE CHARACTERISTICS:
Population: Total number of subjects is 30 -- each subject is own control. "Skin area" is the unit of analysis, thus there are both broccoli sprout extract treated and placebo treated skin areas on each subject (totalling 60 skin areas).
Groups:
- All Participants: Total number of subjects is 30. Each subject will act as his/her own control and receive both treatment and placebo on adjacent skin regions. Thus, 60 skin areas will be randomized.
  Broccoli Sprout Extract: 150 nanomol of sulforaphane/cm2 of skin in 80% acetone for 3 applications on 3 successive days prior to alcohol challenge Placebo Comparator.
Arm/Group | All Participants
Number analyzed (Participants) | 30
Age, Continuous [Mean (Full Range); unit: years] | 34 [25 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 30
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Mean Area of Skin Erythema (Skin Redness)
Description: For three days in a row, volunteers will receive skin treatments with broccoli sprout extract. On day four, their skin will be measured for a baseline skin color reading. Immediately following this reading, the treated areas of the skin will be challenged with 70 percent alcohol and the redness of the skin will again be measured every 30 minutes for the following two hours for skin color changes. The values were collected every 30 minutes after the alcohol skin challenge for 2 hours and were averaged. Mean and 95% Confidence Interval are reported.
Time Frame: mean up to 2 hours
Population: Since experimental conditions were refined part way through the series and only the last 19 individuals' data was deemed suitable for analysis.
Measure: Mean (95% Confidence Interval); unit: centimeters^2
Arm/Group | Broccoli Sprout Extract | Placebo
Number analyzed (Participants) | 19 | 19
centimeters^2 | 3.968 [2.900 to 5.036] | 1.739 [0.912 to 2.567]

ADVERSE EVENTS:
Arm/Group | Broccoli Sprout Extract | Placebo
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 5/30 | 5/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Broccoli Sprout Extract (N=30) | Placebo (N=30)
mild itchy skin or erythema (Skin and subcutaneous tissue disorders) | 5 (5) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes